CLINICAL TRIAL: NCT01054885
Title: A 24-Week Study to Evaluate the Efficacy and Safety of Fluticasone Furoate (FF)/GW642444 Inhalation Powder and the Individual Components Delivered Once Daily (AM) Via a Novel Dry Powder Inhaler Compared With Placebo in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Study of Fluticasone Furoate (FF)/GW642444 Inhalation Powder and the Individual Components in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112207
Record Dates: First submitted 2010-01-14; First posted 2010-01-22 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Efficacy; FEV1; Safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Fluticasone Furoate Inhalation Powder (Experimental): Inhaled Corticosteroid (ICS)
  Interventions: Drug: FF Inhalation Powder
- FF Inhalation Pwdr (Experimental): Inhaled Corticosteroid (ICS)
  Interventions: Drug: FF Inhalation Powder
- Fluticasone Furoate/GW642444 Inhalation Powder (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: FF/GW642444 Inhalation Powder
- FF/GW642444 Inhalation Pwdr (Experimental): Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA)
  Interventions: Drug: FF/GW642444 Inhalation Powder
- GW642444 Inhalation Powder (Experimental): Long Acting Beta Agonist(LABA)
  Interventions: Drug: GW642444 Inhalation Powder
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FF Inhalation Powder — Inhaled Corticosteroid (ICS)
  Arms: FF Inhalation Pwdr; Fluticasone Furoate Inhalation Powder
Drug: FF/GW642444 Inhalation Powder — Inhaled Corticosteroid (ICS)/ Long Acting Beta Agonist(LABA) for COPD
  Arms: FF/GW642444 Inhalation Pwdr; Fluticasone Furoate/GW642444 Inhalation Powder
Drug: GW642444 Inhalation Powder — Long Acting Beta Agonist(LABA)
  Arms: GW642444 Inhalation Powder
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The Purpose of this study is to assess the efficacy and safety of two strengths of the FF/GW642444 Inhalation Powder in subject with Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: outpatient
* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Male or female subjects A female is eligible to enter and participate in the study if she is of:
* Non-child bearing potential OR
* Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods defined in the protocol
* Age: ≥40 years of age at Screening (Visit 1)
* COPD diagnosis: Subjects with a clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [Celli, 2004]
* Tobacco use: Subjects with a current or prior history of ≥10 pack-years of cigarette smoking at Screening (Visit 1).
* Severity of Disease: Subjects with a Screening (Visit 1) measured post-albuterol/salbutamol:
* FEV1/FVC ratio of ≤0.70 and
* FEV1 ≤70% of predicted normal values
* Dyspnea: Achieved a score of ≥2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Screening (Visit 1).

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma
* α1-antitrypsin deficiency: Subjects with α1-antitrypsin deficiency as the underlying cause of COPD
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases, or other active pulmonary diseases
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1)
* Chest X-ray (or CT scan): Subjects with a chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD.
* Hospitalization: Subjects who are hospitalized due to poorly controlled COPD within 12 weeks of Visit 1.
* Poorly controlled COPD: Subjects with poorly controlled COPD, defined as the occurrence of the following in the 6 weeks prior to Visit 1: Acute worsening of COPD that is managed by subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician.
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1.
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular (i.e., pacemaker), neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled.
* Peptic Ulcer disease: Subjects with clinically significant peptic ulcer disease that is uncontrolled.
* Hypertension: Subjects with clinically significant hypertension that is uncontrolled.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
* Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medication or components of the inhalation powder
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol and/or their ipratropium 4 hours prior to spirometry testing at each study visit
* Additional medication: Use of certain medications such as bronchodilators and corticosteroids for the protocol-specified times prior to Visit 1 (the Investigator will discuss the specific medications)
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e., ≤12 hours per day) is not exclusionary.
* Sleep apnea: Subjects with clinically significant sleep apnea who require use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening (Visit 1) or who will enter the acute phase of a Pulmonary Rehabilitation Program during the study.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Prior use of study medication/other investigational drugs
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2009-10-19; Primary Completion 2011-02-01 (Actual); Study Completion 2011-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (116):
- United States (49):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Monterey Park, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Martinez, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, New Tazewell, Tennessee
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (3):
  - GSK Investigational Site, Cipolletti, Río Negro Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Czechia (9):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Tábor
- Germany (13):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Darmstadt, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Japan (10):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Poland (8):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Giżycko
  - GSK Investigational Site, Piekary Śląskie
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Łomża
- Romania (9):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Popeşti-Leordeni
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (8):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Martinez FJ, Boscia J, Feldman G, Scott-Wilson C, Kilbride S, Fabbri L, Crim C, Calverley PM. Fluticasone furoate/vilanterol (100/25; 200/25 mug) improves lung function in COPD: a randomised trial. Respir Med. 2013 Apr;107(4):550-9. doi: 10.1016/j.rmed.2012.12.016. Epub 2013 Jan 16. PMID 23332861
- [Derived] Yang L, Llanos-Paez C, Yang S, Ambery C, Berges A, Kjellsson MC, Karlsson MO. A Combined Model-Based Meta-Analysis of Aggregated and Individual FEV1 Data From Randomized COPD Trials. CPT Pharmacometrics Syst Pharmacol. 2026 Feb;15(2):e70059. doi: 10.1002/psp4.70059. Epub 2025 Jun 19. PMID 40536286
- [Derived] Svedsater H, Dale P, Garrill K, Walker R, Woepse MW. Qualitative assessment of attributes and ease of use of the ELLIPTA dry powder inhaler for delivery of maintenance therapy for asthma and COPD. BMC Pulm Med. 2013 Dec 7;13:72. doi: 10.1186/1471-2466-13-72. PMID 24314123
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112207 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) completed a 2-week single-blind (placebo) Run-in Period (RIP) to assess Baseline rescue use, symptoms, disease stability. Par. were then randomized to a 24-week Treatment Period. A total of 1909 par. were screened, 1577 entered the RIP, of whom 1226 were randomized, 1224 received at least one dose of study medication.
Groups:
- Placebo Run-in: Participants received placebo once daily (OD) in the morning for 2 weeks.
- Placebo: Participants received placebo once daily (OD) in the morning from the dry powder inhaler (DPI) for 24 weeks.
- FF 100 µg OD: Participants received Fluticasone Furoate (FF) 100 micrograms (µg) OD in the morning from the DPI for 24 weeks.
- FF 200 µg OD: Participants received FF 200 µg OD in the morning from the DPI for 24 weeks.
- VI 25 µg OD: Participants received Vilanterol (VI [GW642444]) 25 µg OD in the morning from the DPI for 24 weeks.
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg OD in the morning from the DPI for 24 weeks.
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg OD in the morning from the DPI for 24 weeks.
Period: 2-week, Single-blind Run-In Period
Arm/Group | Placebo Run-in | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Started | 1577 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1226 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 351 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 246 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Closed/Terminated | 68 | 0 | 0 | 0 | 0 | 0 | 0
Period: 24-week, Double-blind Treatment Period
Arm/Group | Placebo Run-in | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Started | 0 | 205 | 204 | 203 | 203 | 204 | 205
Completed | 0 | 146 | 155 | 160 | 161 | 144 | 158
Not Completed | 0 | 59 | 49 | 43 | 42 | 60 | 47
Not completed — Adverse Event | 0 | 18 | 12 | 15 | 15 | 17 | 19
Not completed — Lack of Efficacy-No Sub-Reason | 0 | 0 | 3 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy-Sub-Reason Exacerbation | 0 | 12 | 2 | 5 | 11 | 7 | 7
Not completed — Protocol Violation | 0 | 7 | 7 | 2 | 3 | 8 | 4
Not completed — Protocol Defined Stopping Criteria | 0 | 7 | 12 | 7 | 7 | 15 | 12
Not completed — Study Closed/ Terminated | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 2 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 4 | 1 | 6 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 9 | 7 | 3 | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo OD in the morning from the DPI for 24 weeks.
- FF 100 µg OD: Participants received FF 100 µg OD in the morning from the DPI for 24 weeks.
- VI 25 µg OD: Participants received VI 25 µg OD in the morning from the DPI for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | Total
Number analyzed (Participants) | 205 | 204 | 203 | 203 | 204 | 205 | 1224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.14) | 61.8 (8.28) | 61.8 (9.02) | 61.2 (8.62) | 61.9 (8.79) | 61.1 (8.67) | 61.6 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 52 | 52 | 60 | 68 | 339
  Male | 152 | 150 | 151 | 151 | 144 | 137 | 885
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (HER) | 0 | 2 | 5 | 3 | 4 | 2 | 16
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 2 | 0 | 3
  Japanese/East Asian HER/South East Asian HER | 8 | 5 | 14 | 4 | 8 | 11 | 50
  White | 197 | 197 | 183 | 196 | 190 | 192 | 1155

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean FEV1 Over 0-4 Hours (h) Post-dose at Day 168
Description: Co-Primary Endpoint: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Serial FEV1 measurements were taken electronically by spirometry at BL, weeks 2, 8, 12, and 84 (Day 168). Weighted mean (WM) was calculated using the 0 - 4 h post-dose FEV1 measurements that included the pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits:23 and 24 h after previous morning dose) and post-dose (5, 15, and 30 min and 1, 2, and 4 h) assessments. BL FEV1 is the mean of the two assessments made 30 and 5 min pre-dose at Day 1. WM change from BL was the WM at the visit minus the BL value. Analysis was performed using a repeated measures model with covariates of treatment, smoking status at screening (stratum), BL- mean of the two assessments made 30 and 5 min pre-dose on Day 1, centre grouping, Day, Day by BL and Day by treatment interactions.
Time Frame: Baseline (BL) to Day 168
Population: Intent-to-Treat (ITT) Population: all randomized par. who received at least one dose of study medication. Number of par. presented represent those with data available at the time point being presented; however, all par. in the ITT population without missing covariate information and with at least one post BL measurement are included in the analysis
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 147 | 154 | 162 | 160 | 146 | 158
Liters | -0.012 (0.0189) | 0.034 (0.0187) | 0.029 (0.0185) | 0.173 (0.0184) | 0.202 (0.0190) | 0.197 (0.0184)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.085, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.046, 95% CI 2-sided [-0.006 to 0.098]
Statistical Analysis 2: Comparison: Placebo vs FF 200 µg OD; Test type: Superiority or Other; p = 0.123, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.041, 95% CI 2-sided [-0.011 to 0.093]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.185, 95% CI 2-sided [0.133 to 0.237]
Statistical Analysis 4: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.214, 95% CI 2-sided [0.161 to 0.266]
Statistical Analysis 5: Comparison: Placebo vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.209, 95% CI 2-sided [0.157 to 0.261]
Statistical Analysis 6: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.168, 95% CI 2-sided [0.116 to 0.220]
Statistical Analysis 7: Comparison: FF 200 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.168, 95% CI 2-sided [0.117 to 0.219]
Statistical Analysis 8: Comparison: VI 25 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p = 0.274, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.029, 95% CI 2-sided [-0.023 to 0.081]
Statistical Analysis 9: Comparison: VI 25 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.024, 95% CI 2-sided [-0.027 to 0.075]

2. Primary Outcome: Change From Baseline in Clinic Visit Trough (Pre-bronchodilator and Pre-dose) FEV1 at Day 169
Description: Co-Primary Endpoint: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 7, 14, 28, 56, 84, 112, 140, 168, and 169. BL was defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1.Trough FEV1 was defined as the mean of the FEV1 values obtained 23 and 24 hours after previous morning's dosing. Change from BL was calculated as the average at each visit minus the BL value. Analysis was performed using a repeated measures model with covariates of treatment, smoking status at screening (stratum), BL - mean of the two assessments made 30 minutes pre-dose and immediately pre-dose on Day 1, centre grouping, Day, Day by BL and Day by treatment interactions.
Time Frame: Baseline to Day 169
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 142 | 148 | 155 | 150 | 137 | 153
Liters | 0.004 (0.0189) | 0.048 (0.0187) | 0.012 (0.0185) | 0.103 (0.0185) | 0.148 (0.0191) | 0.135 (0.0185)
Statistical Analysis 1: Comparison: Placebo vs FF 100 µg OD; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.044, 95% CI 2-sided [-0.008 to 0.097]
Statistical Analysis 2: Comparison: Placebo vs FF 200 µg OD; Test type: Superiority or Other; p = 0.756, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.008, 95% CI 2-sided [-0.044 to 0.060]
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.100, 95% CI 2-sided [0.048 to 0.151]
Statistical Analysis 4: Comparison: Placebo vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.144, 95% CI 2-sided [0.091 to 0.197]
Statistical Analysis 5: Comparison: Placebo vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.131, 95% CI 2-sided [0.080 to 0.183]
Statistical Analysis 6: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.100, 95% CI 2-sided [0.047 to 0.152]
Statistical Analysis 7: Comparison: FF 200 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.123, 95% CI 2-sided [0.072 to 0.174]
Statistical Analysis 8: Comparison: VI 25 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p = 0.093, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.045, 95% CI 2-sided [-0.008 to 0.097]
Statistical Analysis 9: Comparison: VI 25 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; p = 0.224, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.032, 95% CI 2-sided [-0.019 to 0.083]

3. Secondary Outcome: Change From Baseline in Chronic Respiratory Disease Questionnaire Self-administered Standardized (CRQ-SAS) Dyspnea Score at Day 168
Description: Considered an 'Other' endpoint by FDA. CRQ-SAS measures 4 domains (mastery, fatigue, emotional function, and dyspnea) of functioning of participants with COPD: mastery (amount of control the participant feels he/she has over COPD symptoms); fatigue (how tired the participant feels); emotional function (how anxious/depressed the participant feels); and dyspnea (how short of breath the participant feels during physical activities). Each domain is measured on a scale of 1-7 (1=maximum impairment; 7=no impairment). Each domain score is calculated separately. Current assessment was done only for dyspnea domain. BL scores are the derived scores for each domain and total at Day 1 pre-dose. Change from BL was calculated as the average at each visit minus the BL value. Analysis performed used a repeated measures model with covariates of treatment, smoking status at screening (stratum), BL (derived scores at Day 1 pre-dose), centre grouping, Day, Day by BL and Day by treatment interactions.
Time Frame: Baseline to Day 168
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 146 | 154 | 161 | 161 | 146 | 156
Scores on a scale | 0.21 (0.077) | 0.10 (0.076) | 0.21 (0.075) | 0.28 (0.075) | 0.45 (0.078) | 0.31 (0.075)

4. Secondary Outcome: Change From Baseline in Peak Post-dose FEV1 (0-4 Hour) on Day 1
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. BL FEV1 is defined as the mean of the assessments made 30 minutes pre-dose and immediately pre-dose on Day 1. If one of these two assessments was missing then BL was defined as the single pre-dose FEV1 value on Day 1. Peak post-dose FEV1 (0-4 hours) is the maximum post-dose FEV1 recorded over the nominal timepoints of 5, 15 and 30 min, 1, 2 and 4 hours post the Day 1 dose. Change from BL is calculated as the peak post-dose FEV1 (0-4 hour) on Day 1 minus BL FEV1. Analysis performed used an Analysis of Covariance (ANCOVA) model with covariates of treatment, smoking status at screening (stratum), BL - mean of the two assessments made 30 minutes pre-dose and immediately pre-dose on Day 1, and centre grouping.
Time Frame: Baseline and Day 1
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of study medication. Only those participants available at the indicated time point and without missing covariate information were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- FVI 25 µg OD: Participants received VI 25 µg OD in the morning from the DPI for 24 weeks.
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | FVI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 204 | 203 | 202 | 201 | 203 | 205
Liters | 0.120 (0.0108) | 0.144 (0.0109) | 0.127 (0.0109) | 0.267 (0.0109) | 0.272 (0.0109) | 0.261 (0.0108)

5. Secondary Outcome: Time to Onset (Increase of 100 Milliliter [mL] From Baseline in 0-4 Hours Post-dose FEV1) on Treatment Day 1
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled from the lungs in one second. Baseline FEV1 is defined as the mean of the two assessments made 30 minutes pre-dose and immediately pre-dose on Day 1. Time to onset on Treatment Day 1 is defined as a 100 mL increase from Baseline in FEV1. Time to increase of 100 mL from Baseline was calculated over the 5, 15, 30 minutes, and 1, 2, and 4 hours time points. A participant who had at least one post-dose FEV1 on Day 1, but did not achieve a 100 mL or more increase from Baseline at any scheduled time-point at which FEV1 was assessed up to and including 4 hours was censored.
Time Frame: Baseline and Day 1
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of study medication. Only those participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 204 | 203 | 202 | 201 | 203 | 205
Minutes | NA [5 to 240] — > 50% of participants were censored; therefore, the median could not be calculated. | 231 [5 to 240] | 242 [5 to 242] | 17 [5 to 240] | 16 [5 to 240] | 17 [5 to 240]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication through the end of treatment (up to Week 24).
Description: An on-treatment AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | Placebo | FF 100 µg OD | FF 200 µg OD | VI 25 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Serious Adverse Events (participants affected / at risk) | 10/205 | 6/204 | 10/203 | 16/203 | 12/204 | 15/205
Other Adverse Events (participants affected / at risk) | 39/205 | 32/204 | 46/203 | 43/203 | 36/204 | 40/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=205) | FF 100 µg OD (N=204) | FF 200 µg OD (N=203) | VI 25 µg OD (N=203) | FF/VI 100/25 µg OD (N=204) | FF/VI 200/25 µg OD (N=205)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 5 | 5 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 3
Infective exacerbation of chronic obstructive airway disease (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=205) | FF 100 µg OD (N=204) | FF 200 µg OD (N=203) | VI 25 µg OD (N=203) | FF/VI 100/25 µg OD (N=204) | FF/VI 200/25 µg OD (N=205)
Nasopharyngitis (Infections and infestations) | 17 | 14 | 20 | 19 | 13 | 13
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 5 | 9 | 8 | 7
Oral candidiasis (Infections and infestations) | 2 | 5 | 5 | 2 | 8 | 4
Oropharyngeal candidiasis (Infections and infestations) | 3 | 0 | 7 | 1 | 3 | 4
Headache (Nervous system disorders) | 15 | 13 | 11 | 20 | 11 | 15
Hypertension (Vascular disorders) | 3 | 3 | 7 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.